CLINICAL TRIAL: NCT01995695
Title: Phase 1 Evaluation of the Safety and Immunogenicity of Live Influenza A Vaccine H7N9 (6-2) AA ca Recombinant (A/Anhui/1/2013 (H7N9) x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H7N9 Disease in the Event of a Pandemic
Brief Title: Safety and Immunogenicity of a Live Attenuated H7N9 Influenza Virus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: URMC 13-001
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Influenza A Virus, H7N9 Subtype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: One Vaccine Dose and One Booster Vaccine Dose (Experimental): Participants will receive one dose of live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine at study entry. They will then receive one dose of inactivated subvirion H7N9 influenza vaccine on Day 98.
  Interventions: Biological: Live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 influenza vaccine
- Group 2: Two Vaccine Doses and One Booster Vaccine Dose (Experimental): Participants will receive two doses of live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine: one dose at study entry and one dose on Day 28. They will then receive one dose of inactivated subvirion H7N9 influenza vaccine on Day 98.
  Interventions: Biological: Live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine; Biological: Inactivated subvirion H7N9 influenza vaccine

INTERVENTIONS:
Biological: Live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine — Participants will receive approximately 10^7.0 focus forming units (FFU) of the live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine. The vaccine will be delivered by an Accuspray nasal spray device (0.25 mL per nostril for a total of 0.5 mL of vaccine).
Biological: Inactivated subvirion H7N9 influenza vaccine — Participants will receive 30 mcg of the inactivated subvirion H7N9 vaccine by intramuscular injection.

SUMMARY:
H7N9 avian influenza (AI) viruses have caused a recent outbreak of severe respiratory disease in humans in China. The purpose of this study is to evaluate the safety and immunogenicity of a live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine in healthy adults. A single dose of inactivated subvirion H7N9 influenza vaccine will be administered 3 months later.

DETAILED DESCRIPTION:
H7N9 AI viruses have recently caused a large outbreak of severe respiratory disease in humans in China. A vaccine for use in the event of an H7N9 AI pandemic is an important research priority. Previous studies have shown that when subjects who received a live bird flu vaccine received a subsequent "booster" dose of inactivated bird flu vaccine, a vigorous antibody response was detected. The inactivated vaccine served as a way to probe the immune response to the initial live vaccine. The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of a live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine in healthy adults, and to administer a booster dose of an inactivated subvirion H7N9 influenza vaccine 3 months later.

This study will enroll healthy adults who are willing to remain in an isolation unit in an inpatient clinic for several days during the study. They will be randomly assigned to receive either one dose (Group 1) or two doses (Group 2) of the live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine, which will be delivered by a nasal spray device. Participants in both groups will receive one "booster" dose of inactivated subvirion H7N9 influenza vaccine 3 months later in an outpatient setting. All participants will be admitted to the inpatient clinic and will receive one dose of the live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine 2 days after entering the clinic. Participants will remain in the inpatient clinic for approximately 9 days after receiving the vaccine. While in the clinic, participants will undergo medical history reviews, blood collections, urine collections, physical examinations, nasal wash procedures, and vital sign measurements.

Participants in Group 1 will attend a study visit at Day 28 and undergo a medical history review, blood collection, and a nasal wash. Participants in Group 2 will be readmitted to the inpatient clinic 2 days prior to receiving a second dose of the live attenuated H7N9 A/Anhui/13 ca influenza virus vaccine at Day 28. They will remain in the clinic for approximately 9 days after receiving the vaccine; while in the clinic, they will take part in the same study procedures as during the first inpatient visit.

All participants will attend a study visit at Day 56 and undergo a medical history review, blood collection, and a nasal wash. At Day 98, all participants will receive one "booster" dose of the inactivated subvirion H7N9 influenza vaccine, as outpatients. They will attend additional study visits on Days 101, 105, 112, 126, 154, and 180, which may include medical history reviews; physical examinations; and urine, blood, and nasal secretion collections.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 years and 49 years of age, inclusive. Children will not be recruited or enrolled in this study because they are not in the apparent risk group, and for safety considerations and because of the need for isolation.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Agree to storage of blood specimens for future research
* Available for the duration of the trial
* Willingness to participate in the study as evidenced by signing the informed consent document
* Female participants of child-bearing potential must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse; surgical sterilization). All female participants will be considered being of child-bearing potential except those who have undergone hysterectomy and those in whom menopause occurred at least 1 year prior to the study.

Exclusion Criteria:

* Pregnancy, as determined by a positive human choriogonadotropin (beta-HCG) test
* Currently breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing. Alanine aminotransferase (ALT) levels greater than two times the upper normal limit will be exclusionary at baseline, prior to vaccination.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Previous enrollment in an H7 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N9 influenza A virus (serum HAI titer greater than 1:8)
* Positive urine drug toxicology test indicating narcotic use/dependency
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis
* Allergy to oseltamivir as determined by participant report
* Current diagnosis of asthma or reactive airway disease (within the past 2 years)
* History of Guillain-Barré Syndrome
* Positive ELISA and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1)
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* History of asplenia
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study:

  * A current smoker includes anyone stating they currently smoke any amount of a tobacco product.
  * The decision to exclude a potential participant is determined by medical history and a clinician's clinical judgment based on the physical examination.
  * After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Travel to the Southern Hemisphere within 14 days prior to study vaccination
* Travel on a cruise ship within 14 days prior to study vaccination
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events that occur during the acute monitoring (inpatient) phase of the study | Measured through Day 9 (Group 1) or Day 37 (Group 2)
Area under the curve (AUC) of nasal virus shedding after each dose of vaccine, as assessed by liquid titration of nasal secretions on Madin Darby canine kidney (MDCK) cells at 33°C | Measured through Day 180
Vaccine virus shedding on one or more days on Days 2 through 9 as assessed by culture or real-time reverse transcriptase polymerase chain reaction (rRT-PCR) | Measured through Day 9
Evidence of a 4-fold or greater increase in either hemagglutination inhibition (HAI) or microneutralization (MN) antibody comparing pre-vaccination to either Day 29 or Day 56 post-dose two samples | Measured through Day 56
Development of serum antibody assessed by either HAI or MN assays | Measured through Day 180

SECONDARY OUTCOMES:
Development of a significant increase in nasal secretion HA-specific antibody assessed by enzyme-linked immunosorbent assay (ELISA) | Measured through Day 180
Development of greater than 200 influenza-specific interferon-gamma-secreting cells per million lymphocytes as assessed by enzyme-linked immunosorbent spot (ELISPOT) on Day 28 after immunization | Measured through Day 28
Detection of influenza-specific immunoglobulin G (IgG) or IgA secreting B cells on Day 7 following vaccination assessed by antibody secreting cells (ASC) assay | Measured through Day 7

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Sobhanie M, Matsuoka Y, Jegaskanda S, Fitzgerald T, Mallory R, Chen Z, Luke C, Treanor J, Subbarao K. Evaluation of the Safety and Immunogenicity of a Candidate Pandemic Live Attenuated Influenza Vaccine (pLAIV) Against Influenza A(H7N9). J Infect Dis. 2016 Mar 15;213(6):922-9. doi: 10.1093/infdis/jiv526. Epub 2015 Dec 9. PMID 26655841